CLINICAL TRIAL: NCT03145935
Title: Diagnosis Accuracy of Abdominal Compression and Hemoconcentration to Detect Diuretic Induced Fluid Removal Intolerance.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hopital Louis Pradel (Other)
Responsible Party: Principal Investigator, Matthias Jacquet-Lagrèze, Medical doctor, Principal investigator, Hopital Louis Pradel
Other Study IDs: ANSM 2017-A01334-49.
Record Dates: First submitted 2017-05-05; First posted 2017-05-09 (Actual); Last update posted 2019-04-12 (Actual); Status verified 2019-04

CONDITIONS: Hypovolemia; Diuretic Toxicity; Fluid Overload
MeSH Terms: conditions — Hypovolemia; Edema | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Abdominal compression (AC) — An echocardiography with stroke volume measurement coupled with an abdominal compression will be performed before and after ta diuretics induced diuresis of 10ml/kg in pediatric patients hospitalized in a pediatric intensive care unit (PICU) diagnosed with fluid overload
  Other Names: Echocardiographic assessement of volume status
Diagnostic Test: blood sample — proteinemia and hematocrit will be measured before and after a diuretics induced diuresis of 10ml/kg

SUMMARY:
Fluid overload increases morbidity and mortality of pediatrics patients in intensive care unit (ICU). It could be interesting to predict the decrease in stroke volume when diuretics are prescribed. Nevertheless, no test predict a decrease of stroke volume in a context of a diuretics induced depletion. Abdominal compression (AC) coupled with echocardiographic measurement of the stroke volume can predict fluid responsiveness and is a good tool to assess preload dependency. Another point is that during depletion refilling can occur. We aim to assess the diagnostic accuracy of abdominal compression to predict a decrease of the stroke volume of 15 % during diuretic-induced depletion of 10 ml/kg of diuresis. Secondary outcome will assess the hemoconcentration during depletion to diagnose a decrease of stroke volume during diuretic induced depletion

DETAILED DESCRIPTION:
Fluid overload increases morbidity and mortality of pediatrics patients in intensive care unit (ICU). The pediatric intensivist has a priority to decrease unnecessary fluid load and to make the fluid balance negative in case of fluid overload. Diuretics help to make the fluid balance negative but can lead to a reduction of volemia that can lead to hypovolemia. Hypovolemia can induce a reduction of stroke volume and cardiac index that can alter tissue perfusion and increase organ dysfunction.

It could be interesting to predict the decrease in stroke volume when diuretics are prescribed. Nevertheless, no test predict a decrease of stroke volume in a context of a diuretics induced depletion.

The concept of preload dependency described by frank-starling is interesting in that context.

Preload dependency is a state of the working heart characterized by a modification of stroke volume when a modification of preload is done. Conversely, no preload dependency is a state of the working heart characterized by no modification of stroke volume when a modification of preload is done.

If the heart is in a state of preload dependency, a reduction of preload induced by diuretics depletion might induce a reduction of stroke volume. Conversely, if the heart is in a state of no preload dependency a reduction of preload induced by a diuretics depletion might not induce a reduction of stroke volume Abdominal compression coupled with echocardiographic measurement of the stroke volume can predict fluid responsiveness and is a good tool to assess preload dependency.

Another point is that during depletion refilling can occur. Studies performed during hemodialysis have shown that refilling maintains a stable hematocrit during depletion. the absence of refilling is characterized by an hemoconcentration

We aim to assess the diagnostic accuracy of abdominal compression to predict a decrease of the stroke volume of 15 % during diuretic induced depletion of 10ml/kg of diuresis. Secondary outcome will assess the hemoconcentration during depletion to diagnose a decrease of stroke volume during diuretic induced depletion

ELIGIBILITY:
Inclusion Criteria:

* Height year old or less
* Patient hospitalized in the pediatric intensive care unit of the investigation center.

presenting symptoms of fluid overload characterized with:

* Peripheral edema.
* An increase of 10% between the first day in ICU and inclusion date

  * the attending physician should have decided to evaluate hemodynamic with iterative echocardiography
  * the attending physician, who is not the investigator has decided to administer diuretics

Exclusion Criteria:

* Patient or Holder of parental authority refusal to participate
* Dehydration with natremia over 150 mmol/L or clinical signs of dehydration
* Suspected abdominal hypertension
* recent abdominal surgery with abdominal pain induced by abdominal examination.

Max Age: 8 Years | Sex: All
Age Groups: Child
Study Population: Pediatric patients under 8 years old, hospitalized in the pediatric intensive care unit of investigation center.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2017-05-10 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Stroke volume index (SVi) variation induced by abdominal compression ΔSVi-AC | 2 hours
  Variation of stroke volume index measured with echocardiography induced by abdominal compression. We will test if stroke volume index variation during abdominal compression can predict a decrease of 15 % of the stroke volume during a 10 ml/kg diuresis induced by diuretics administration.

SECONDARY OUTCOMES:
Hemoconcentration with protides | 2 hours
  proteinemia variation. We will test if proteinemia variation can predict a diagnose a reduction of 15 % of the stroke volume during a 10 ml/kg diuresis induced by diuretics administration.
Hemoconcentration with hematocrit | 2 hours
  Hematocrit variation. We will test if hematocrit variation can predict a diagnose a reduction of 15 % of the stroke volume during a 10 ml/kg diuresis induced by diuretics administration.
Respiratory variation of the maximum aortic velocity of the left ventricular outflow tractΔVpeak | 2 hours
  Variation of the maximum velocity of the left ventricular outflow tract induced by ventilation. We will test if ΔVpeak can predict a decrease of 15 % of the stroke volume during a 10 ml/kg diuresis induced by diuretics administration.
Respiratory variation of the inferior vena cava diameter ΔIVC | 2 hours
  Variation of inferior vena cava diameter induced by ventilation. We will test if ΔIVC can predict a decrease of 15 % of the stroke volume during a 10 ml/kg diuresis induced by diuretics administration.

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Louis Pradel, Bron, Auvergne-Rhône-Alpes, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Foland JA, Fortenberry JD, Warshaw BL, Pettignano R, Merritt RK, Heard ML, Rogers K, Reid C, Tanner AJ, Easley KA. Fluid overload before continuous hemofiltration and survival in critically ill children: a retrospective analysis. Crit Care Med. 2004 Aug;32(8):1771-6. doi: 10.1097/01.ccm.0000132897.52737.49. PMID 15286557
- [Result] Sinitsky L, Walls D, Nadel S, Inwald DP. Fluid overload at 48 hours is associated with respiratory morbidity but not mortality in a general PICU: retrospective cohort study. Pediatr Crit Care Med. 2015 Mar;16(3):205-9. doi: 10.1097/PCC.0000000000000318. PMID 25581632
- [Result] Li Y, Wang J, Bai Z, Chen J, Wang X, Pan J, Li X, Feng X. Early fluid overload is associated with acute kidney injury and PICU mortality in critically ill children. Eur J Pediatr. 2016 Jan;175(1):39-48. doi: 10.1007/s00431-015-2592-7. Epub 2015 Jul 24. PMID 26206387
- [Result] Monnet X, Cipriani F, Camous L, Sentenac P, Dres M, Krastinova E, Anguel N, Richard C, Teboul JL. The passive leg raising test to guide fluid removal in critically ill patients. Ann Intensive Care. 2016 Dec;6(1):46. doi: 10.1186/s13613-016-0149-1. Epub 2016 May 20. PMID 27207178